CLINICAL TRIAL: NCT05804149
Title: Effect of Acupuncture and Low Caloric Diet on Primary Hypothyroidism and Irregular Menstruation in Infertile Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Sedky, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: No:P.T.REC/012/002825
Record Dates: First submitted 2023-02-16; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Primary Hypothyroidism; Acupuncture; Irregular Menstruation; PCO
Keywords: primary hypothyroidism; acupuncture; low caloric diet; infertile women
MeSH Terms: conditions — Hypothyroidism; Menstruation Disturbances | interventions — Acupuncture Therapy; Thyroxine; Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Each woman in both groups (control and study) will receive thyroxine tablets (levothyroxine) (1tablet per day) describe by the physician. Levothyroxine is usually taken 30-60 minutes before breakfast, or four hours after food, as certain substance such as food and calcium can inhabit the absorption of levothyroxine Acupuncture will be applied with a total duration of 35-45 minutes, 2 sessions per week for 4 months.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Each patient in the study group will be instructed about the beneficial effect of the acupuncture.
  * Each woman in the study group will assume side lying position with uncovered treatment area,
  * thyroxine tablets (levothyroxine) (1tablet per day) describe by the physician. Levothyroxine is usually taken 30-60 minutes before breakfast, or four hours after food, as certain substance such as food and calcium can inhabit the absorption of levothyroxine.
  * low caloric diet regime consisting of 1200 to 800Kcal/ day for 4 months.
  * Fine sterile needles will be used with a size 0.25x25mm. They will be inserted to various depths (2-5 cm) at acupoints points on the body according to site and fat deposition. 16 needles will be used in the treatment
  Interventions: Device: acupuncture; Drug: Thyroxine; Dietary Supplement: low caloric diet
- control group (Other): Each woman in both groups (control and study) will receive thyroxine tablets (levothyroxine) (1tablet per day) describe by the physician. Levothyroxine is usually taken 30-60 minutes before breakfast, or four hours after food, as certain substance such as food and calcium can inhabit the absorption of levothyroxine Each woman in both groups will follow a low caloric diet regime consisting of 1200 to 800Kcal/ day for 4 months. The regime will start with 1200 Kcal for the first month and 1100 for the second month then 900 Kcal for the third month until reach 800 Kcal in fourth month.
  Interventions: Drug: Thyroxine; Dietary Supplement: low caloric diet

INTERVENTIONS:
Device: acupuncture — study group take acupuncture Acupuncture was applied with a total duration of 35-45 minutes, 2 sessions per week for 4 months.
  Arms: study group
Drug: Thyroxine — Each woman in both groups (control and study) will receive thyroxine tablets (levothyroxine) (1tablet per day) describe by the physician. Levothyroxine is usually taken 30-60 minutes before breakfast, or four hours after food, as certain substance such as food and calcium can inhabit the absorption of levothyroxine
  Other Names: levothyroxine
Dietary Supplement: low caloric diet — Each woman in both groups will follow a low caloric diet regime consisting of 1200 to 800Kcal/ day for 4 months. The regime will start with 1200 Kcal for the first month and 1100 for the second month then 900 Kcal for the third month until reach 800 Kcal in fourth month.

SUMMARY:
the goal of this randomize clinical trial is to compare in 60 infertile women with hypothyroidism. selected from national Nutritional institute out clinic. the main question it aims to answer is:

• There an effect of acupuncture and low caloric diet on primary hypothyroidism and irregular menstruation in infertile women.

all participants were received• thyroxine tablets (levothyroxine) • a low caloric diet regime.

researchers compared study group (30 infertile women with hypothyroidism) to see the effect of acupuncture sections on hypothyroidism.

DETAILED DESCRIPTION:
Each woman was instructed carefully about the assessment and treatment procedures and a consent form has been signed by each woman before starting of this study,

* Each patient in the study group was instructed about the beneficial effect of the Acupuncture.
* Each woman in the study group assumed supine position for the points (DU20, GB20, ST9, LI4, RN6, RN4, SP9, ST36, SP6, KI3, LR2). and prone position for DU14, BL15, BL20, BL23, DU4 with uncovered treatment area, which was cleaned with alcohol and hair was removed.

Acupuncture was applied on a room temperature of 37. Fine sterile needles used with a size 0.25x25mm. They were inserted to various depths (2-5 cm) at acupoints points on the body according to site and fat deposition. 16 needles were used in the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sixty PCOS women will be evaluated for presence of hirsutism, acne, irregular menses. They will be diagnosed for presence of cysts by Ultrasonography apparatus.
* They will complain from primary hypothyroidism. Their thyroid-stimulating hormone (TSH) will be >4.0mu/l and free tetraiodothyronine (FT4) will be <0.8ng/dl.
* Their luteinizing hormone / follicle-stimulating hormone (LH/FSH) ratio will be <1.
* Their age will range from 20-35 years old.
* Their body mass index (BMI) will be > 25 kg/m2 and < 39.9 kg/m2.

Exclusion Criteria:

* History of previous neurological disorders, previous thyroidectomy, and surgical removal of uterus.
* Presence of hemorrhage, carcinoma, metal implants and using of immune suppressant drugs.
* Presence of endometriosis, uterine fibroids, primary ovary insufficiency, fallopian tube damage or blockage, pelvic adhesion, autoimmune disorders, implantation failure, and infections.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2023-02-12 (Actual)

PRIMARY OUTCOMES:
Thyroid hormones (TSH). (mu/l) | change from TSH at 4 months.
  60 participants with hypothyroidism assessed by blood analysis for thyroid hormones to measure percentage of improvement of hypothyroidism. ELISA plate reader used to measure thyroid hormones including (TSH) measured by mu/l, before starting and after the end of the study course.
Thyroid hormones (FT4). (ng/dl) | change from FT4 at 4 months.
  60 participants with hypothyroidism assessed by blood analysis for thyroid hormones to measure percentage of improvement of hypothyroidism. ELISA plate reader used to measure thyroid hormones including (FT4) measured by ng/dl, before starting and after the end of the study course.
BMI (kg/m2). | change from BMI at 4 months.
  60 infertile women with hypothyroidism assessed by Weight-Height scale. to measure weight (kg) and height (cm) to calculate BMI at starting and after the end of the study course. BMI will be calculated according to the formula: BMI=Weight/Height square (kg/m2).
reproductive hormones including LH(IU/L) | change LH at 4 months.
  60 participants with hypothyroidism assessed by blood analysis for reproductive hormones to measure percentage of improvement of infertility (PCOS). ELISA plate reader used to measure (LH) measured by (IU/L) before starting and after the end of the study course.
FSH (mIU/mL) | change from FSH at 4 months.
  60 participants with hypothyroidism assessed by blood analysis for reproductive hormones to measure percentage of improvement of infertility (PCOS). ELISA plate reader used to measure (FSH) measured by (mIU/mL), before starting and after the end of the study course.
Health-Related Quality-of-Life (PCOS Questionnaire) (score from 26:182 units on scale) | change from PCOS Questionnaire at 4 months.
  60 participants infertile women assessed by Health-Related Quality-of-Life Questionnaire (PCOSQ) to asses health and health related quality of life issues including emotion, body hair, weight, infertility problems, and menstrual problems for each woman in both control and study groups before starting and after the end of the study course. Score from 26:182 units on scale as questionnaire consists of 26 questions, foreach question, there is seven rating options. heigh score means more improvement, while low score means less improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Eman Sedky, Cairo, Maadi, Egypt

IPD SHARING:
Plan to Share IPD: No